CLINICAL TRIAL: NCT01507727
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled (Standard Therapy + Placebo) Study to Evaluate the Efficacy and Safety of the Tolvaptan Tablets in Patients With Non-hypovolemic Non-acute Hyponatremia
Brief Title: Efficacy and Safety Study of the Tolvaptan Tablets in Patients With Non-hypovolemic Non-acute Hyponatremia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Beijing 302 Hospital (Other); Beijing Anzhen Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HENGRUI20111231
Record Dates: First submitted 2012-01-05; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Non-hypovolemic Non-acute Hyponatremia
Keywords: hyponatremia; Non-hypovolemic and Non-acute hyponatremia; Tolvaptan
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Tolvaptan (Experimental)
  Interventions: Drug: Tolvaptan
- Drug: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Tablet;15mg/tab; 30mg/tab; 15/30/60mg/day for 7 days Plus conventional therapy according to each patient's underlying disease, such as CHF, hepatic cirrhosis and SIADH or others.
  Arms: Drug: Tolvaptan
Drug: Placebo — placebo plus conventional therapy according to each patient's underlying disease, such as CHF, hepatic cirrhosis and SIADH or others.
  Arms: Drug: Placebo

SUMMARY:
This drug has been developed to treat Hyponatremia. The primary purpose of this study is to verify the efficacy and safety of seven-day repeated oral administration of tolvaptan at 15, 30, and 60 mg or placebo in patients with Non-hypovolemic Non-acute Hyponatremia secondary to Congestive Heart Failure (CHF), hepatic cirrhosis or Syndrome of Inappropriate Antidiuretic Hormone (SIADH), despite receiving standard therapy. This study is being conducted in China.

ELIGIBILITY:
Inclusion Criteria (for CHF):

1. Patients with CHF who exhibit edema, jugular venous distention, hepatomegaly, or pulmonary congestion.
2. Non-hypovolemic and Non-acute hyponatremia with a serum sodium < 135mEq/L before randomization.
3. Patients who have taken furosemide at 40 mg/d or more (oral dosing) without alteration of dosage for the 3 days of the observation period.
4. Patients whose body weight has been stable (±1.0 kg) for 2 days prior to commencement of study drug administration.
5. Age:18～80 (when informed consent is obtained)，male or female.
6. In-patient subjects.
7. Informed consent.

Inclusion Criteria (for hepatic cirrhosis):

1. Patients with hepatic edema.
2. Non-hypovolemic and non acute hyponatremia with a serum sodium < 135mEq/L before randomization.
3. Age:18～65 (when informed consent is obtained)，male or female.
4. In-patient subjects.
5. Informed consent.

Inclusion Criteria (for SIADH and others):

1. Patients with SIADH arising from a variety of etiologies.
2. Non-hypovolemic and non acute hyponatremia with a serum sodium < 135mEq/L before randomization.
3. Age:18～80 (when informed consent is obtained)，male or female.
4. In-patient subjects.
5. Informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The change of average daily Area Under the Curve (AUC) of serum sodium by day 4 and 7 comparing with baseline serum sodium level within the double-blind therapy period | 4 and 7 days

SECONDARY OUTCOMES:
Percentage of patients with normalized serum sodium at Day 4 | 4 day
Percentage of patients with normalized serum sodium at Day 7 | 7 day
Time to first normalization in serum sodium | up to 7 days
Change from baseline in serum sodium at Day 4 | 4 day
Change from baseline in serum sodium at Day 7 | 7 day
Percentage of patients requiring fluid restriction at any time during the double-blind therapy period of the study | up to 7 days
24-hour urine output | day 1, day 2, day 3, day 4, day 5, day 6 and day 7
Change from baseline in body weight (hypervolemic patients only) | day 1, day 2, day 3, day 4, day 5, day 6 and day 7
Fluid balance (hypervolemic patients only) | day 1, day 2, day 3, day 4, day 5, day 6 and day 7
The percentage of patients who are designated as treatment failure due to the need for saline infusion, with or without fluid restriction | up to 7 days
For CHF patients, improvement of symptoms and relevant physical examination measures | day 1, day 2, day 3, day 4, day 5, day 6 and day 7
For hepatic edema patients, improvement of symptoms and relevant physical examination measures or ultrasound test findings | day 1, day 2, day 3, day 4, day 5, day 6 and day 7

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cardiology, Beijing An Zhen Hospital Affiliated to Capital University of Medical Science, Beijing
  - Endocrinology, Beijing Friendship Hospital, Beijing
  - Hepatology, No. 302 Hospital, Beijing